CLINICAL TRIAL: NCT06708702
Title: Phase II Study to Evaluate the Effectiviness of copaíba-based Mouthwash in Oral Mucotitis Prevention and Treatment in Oral Cancer Patients During Radioteraphy
Brief Title: Copaíba-based Mouthwash in Oral Mucotitis Prevention and Treatment in Oral Cancer Patients During Radioteraphy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto Nacional de Cancer, Brazil (Other Government)
Responsible Party: Principal Investigator, Heliton Spindola Antunes, PhD, Instituto Nacional de Cancer, Brazil
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 76178323.4.0000.5274
Record Dates: First submitted 2024-11-05; First posted 2024-11-27 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Oral Mucositis; Oral Mucositis (Ulcerative) Due to Radiation; Oral Mucositis (Ulcerative) Due to Antineoplastic Therapy; Oral Mucositis Due to Radiation
Keywords: oral mucositis; radiotheraphy; copaiba; low power laser theraphy
MeSH Terms: conditions — Stomatitis; Ulcer

STUDY DESIGN:
Intervention Model Description: This is a phase II, randomized, placebo-controlled, double-blind study in a single institution, to evaluate the effectiveness of copaiba-based mouthwash in preventing oral mucositis in the tumor area in patients with oral cancer undergoing RT alone or in combination with CT. The participant will be randomized 1:1 to the study groups in a stratified manner according to the oncological treatments to which the patient will be subjected, according to the groups: exclusive treatment with RT and treatment with RT associated with CT. Randomization will be carried out using the REDCap® program by a non-blinded pharmacist, trained for this role.
  Participants' daily care (outcome assessment) will begin on the first day of RT, and continue until the end of it, regardless of whether the patient has already reached the study's primary outcome or not.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be blind to the group in which they are included, as will the study team. The non-blind team will be composed of the pharmacy team, that will be responsabli for the randomization and for dispensing of the investigational product/placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Copaíba (Experimental)
  Interventions: Drug: Copaíba mouthwash
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo mouthwash

INTERVENTIONS:
Drug: Copaíba mouthwash — A 15% aqueous solution of copaíba (Copaifera Officinalis Resin) manufactured by Interativo Farmácia de Manipulação will be used, under the formula of copaíba oil (Copaifera Officinalis Resin) 15%, liquid mint aroma 5%, tween 80 1%, aqueous solution (Distilled water + Nipagin 0.1%) qsp 100%.
  Patients will receive the solution once a week. They will be instructed to shake the bottle before use for homogenization, to use 10mL of the solution for each mouthwash (which should be measured in the 10mL measuring cup that comes with each bottle), 4 times a day, rinsing vigorously for 1 minute and discarding all the solution after use.
  Arms: Copaíba
Drug: Placebo mouthwash — Placebo will be used, under the formula of liquid mint flavor 5%, Nipagim 0.1%, and distilled water qsp 60 ml, packed in packaging compatible with that of the product under investigation, maintaining the same physical characteristics to maintain blinding. The product will be stored at room temperature and stored in the INCA pharmacy.
  Patients will receive the solution once a week. They will be instructed to shake the bottle before use for homogenization, to use 10mL of the solution for each mouthwash (which should be measured in the 10mL measuring cup that comes with each bottle), 4 times a day, rinsing vigorously for 1 minute and discarding all the solution after use.
  Arms: Placebo

SUMMARY:
Oral mucositis is the most significant acute toxicity of oral cavity radiotherapy. The available scientific evidence supports its preventive and therapeutic approach with low-level laser; however, this is unsuitable for tumor regions due to the risk of stimulating cellular metabolism. In this sense, an alternative treatment becomes necessary. Based on the preliminary results of the phase I study, a double-blind, randomized phase II study is suggested to evaluate the effectiveness of copaiba-based mouthwash in the prevention of oral mucositis in patients undergoing radiotherapy for oral cavity tumors. Patients will be randomized into 2 groups: A (copaíba) and B (placebo) and will use the mouthwash 4x/day. Each group will have 20 patients and be blind to the group in which they are included. They will be evaluated daily by a dental surgeon about oral mucositis, pain in the oral cavity and oropharynx, and dysphagia and will undergo daily laser therapy sessions, until the end of radiotherapy.

DETAILED DESCRIPTION:
Oral cavity cancer represents the 8th most common type in Brazil, with an estimated 15,100 new cases for each year of the 2023-2025 period. It depends on the patient's clinical condition, tumor location, and staging, involving surgery, chemotherapy (CT), or radiotherapy (RT), alone or in combination. RT involves doses between 50 and 70 Gy and, in addition to the action on the tumor, it produces toxicity in adjacent tissues, compromising the patient's quality of life.

Oral mucositis (OM) is the most significant acute toxicity related to RT associated or not with CT for tumors in this location.7,8 Its preventive and therapeutic approach has been proposed in several ways, but for RT of oral cavity tumors, it has There is evidence for the use of low-level laser therapy (LBP) and benzydamine hydrochloride. However, benzydamine hydrochloride is effective for those who received RT doses of up to 50 Gy, and the application of LBP in the tumor region is contraindicated as its effect is due to the activation of receptors of the respiratory chain, causing stimulation of cellular metabolism. Therefore, OM conditions tend to be severe in these locations, especially in patients with oral tumor lesions. In this sense, the need for an auxiliary treatment method becomes evident.

A phase I study with copaiba (CPB) in patients with oral cancer undergoing RT was previously developed by this group. In this case, the use of the mouthwash did not trigger dose-limiting toxicity in any of the treated patients, allowing us to conclude that the maximum tested dose of 15% used 4 times/day is safe for the development of a phase II study. None of the patients reported pain or burning related to the use of mouthwash in the absence of OM lesions, suggesting that it is safe and non-toxic for this use. The preliminary assessment of the effectiveness of the mouthwash showed the occurrence of OM lesions in 89.5% of patients, at most grade 3; None of the patients evaluated developed grade 4 mucositis lesions according to the WHO scale. None of the patients evaluated in the study needed to interrupt RT or QT due to OM injuries.

OBJECTIVES Main objective: to evaluate the effectiveness of copaiba-based mouthwash in preventing and treating oral mucositis in patients with oral cancer undergoing radiotherapy.

Secondary objectives: evaluate the safety of copaiba mouthwash in patients who use it; compare the incidence of oral mucositis in tumor and non-tumor areas in the two groups; compare the oral cavity pain index in the two groups; compare the oropharyngeal pain index in the two groups; compare the dysphagia index in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older;
* Patients enrolled at INCA diagnosed with malignant neoplasms located in the oral cavity or oropharynx with an extension of the lesion to the oral cavity (IDC-10 C01 to C06 or IDC10); with the indication of exclusive RT (using the Intensity Modulated Radiotherapy (IMRT)/ Volumetric Modulated Arcotherapy (VMAT) technique) or combined with surgery and/or CT;
* Patients with expected RT doses between 50 and 70Gy;
* Patients capable of understanding and adhering to the protocol;
* Patients capable of performing the oral hygiene protocol;
* Patients who, after the information and instructions, can provide the free and informed consent form.

Exclusion Criteria:

* Patients who are receiving drugs for the treatment and/or prevention of OM;
* Patients undergoing RT with planning that excludes the oral cavity from the irradiation field;
* Patients who report any allergy to CPB-based compounds.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Oral mucositis ulcers in tumoral area | From date of randomization until the date of first documented ulcer or date of last RT session/ mouthwash use day, whichever came first, assessed up to 7 weeks
  To evaluate the incidence of oral mucositis (ulcers) in the tumor area in patients with oral cancer undergoing radiotherapy using copaiba-based mouthwash

SECONDARY OUTCOMES:
Mouthwashs safety | From date of randomization until the date of last RT session/ mouthwash use day, assessed up to 7 weeks
  Assess the safety of copaiba mouthwash/placebo
Oral Mucositis (OMS) | From date of randomization until the date of last RT session/ mouthwash use day, assessed up to 7 weeks
  Compare the incidence of maximum grade (grade 1, 2, 3, or 4 according to the WHO scale) of oral mucositis between the two groups
Oral Mucositis ulcers (Sonis) | From date of randomization until the date of last RT session/ mouthwash use day, assessed up to 7 weeks
  Compare the average ulcerated area in the tumor area between the two groups according to the Sonis scale
Oral Mucositis erithema (Sonis) | From date of randomization until the date of last RT session/ mouthwash use day, assessed up to 7 weeks
  Compare the average area with erythema in the tumor area between the two groups according to the Sonis scale
Oral Mucositis (Sonis) | From date of randomization until the date of last RT session/ mouthwash use day, assessed up to 7 weeks
  Compare the average sum of the ulcerated area with the area of erythema in the tumor area between the two groups according to the Sonis scale
Oral pain | From date of randomization until the date of last RT session/ mouthwash use day, assessed up to 7 weeks
  Compare the oral cavity pain index in the two groups according to the VAS and the CTCAE v5.0
Oropharingeal pain | From date of randomization until the date of last RT session/ mouthwash use day, assessed up to 7 weeks
  Compare the oropharyngeal pain index in the two groups according to the VAS and CTCAE v5.0
Dysphagia | From date of randomization until the date of last RT session/ mouthwash use day, assessed up to 7 weeks
  Compare the dysphagia index in the two groups according to CTCAE v5.0
Siamoletry | At first RT day/ mouthwash use day, in the midle of the RT sessions/ mouthwash use and at last RT session/ mouthwash use day, assessed up to 7 weeks
  Compare unstimulated sialometry values in the two groups at the beginning, middle, and end of treatment
Cytokines | At first RT day/ mouthwash use day, in the midle of the RT sessions/ mouthwash use and at last RT session/ mouthwash use day, assessed up to 7 weeks
  Compare the levels of pro-inflammatory cytokines IL-1 β, IL-6, and TNF- α in the two groups at the beginning, middle, and end of treatment

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Instituto Nacional de Cancer, Brazil, Rio de Janeiro, Rio de Janeiro
  - Instituto Nacional de Cancer, Rio de Janeiro, Rio de Janeiro

IPD SHARING:
Plan to Share IPD: No